CLINICAL TRIAL: NCT03455387
Title: Evaluation of the Serum Markers sFLt1 and PlGF for the Prediction of the Complications of the Placental Vascular Pathologies in the 3rd Quarter of the Pregnancy.
Acronym: PRECOPE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Metropole Savoie (Other)
Responsible Party: Sponsor
Other Study IDs: CHMS16001
Record Dates: First submitted 2018-02-28; First posted 2018-03-06 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Pre-Eclampsia; HELLP Syndrome; Fetal Death; Eclampsia; Placental Abruption; Fetal Growth Retardation, Antenatal
Keywords: sFLt1; PlGF
MeSH Terms: conditions — Pre-Eclampsia; HELLP Syndrome; Fetal Death; Eclampsia; Abruptio Placentae; Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- sampling of serum marker Flt1 and PIGF: sampling of the serum markers sFlt1 and PlGF , every 3 days,until delivery
  Interventions: Diagnostic Test: sampling of the serum marker sFlt1 and PlGF

INTERVENTIONS:
Diagnostic Test: sampling of the serum marker sFlt1 and PlGF — sampling of the serum markers sFlt1 and PlGF , every 3 days,until delivery

SUMMARY:
The pre-eclampsia is a frequent pathology, concerning approximately 5 % of the pregnancies.The pre-eclampsia can evolve into severe maternal and\or foetal complications and is a major cause of mortality.

The purpose of the study will to estimate the relevance of the serum markers sFlt1 and PlGF to predict the arisen of severe complications at these patients, what would allow to decrease the materno-fœtale morbi-mortality due to the pathology.

DETAILED DESCRIPTION:
The pre-eclampsia is a frequent pathology, concerning approximately 5 % of the pregnancies. It is a major cause of mortality, mainly in the developing country. His incidence tends to increase in the developed countries. In the absence of adapted coverage, the pre-eclampsia can evolve into severe maternal and\or foetal complications (eclampsia, foetal intra-uterine, dead HELLP syndrome, lung acute oedema, stunting in utero).

The pre-eclampsia is a part of placental vascular pathologies. Several studies showed that these pathologies are due to a defect of trophoblastic invasion, secondary in an imbalance in the balance of factors pro and antiangiogéniques (PlGF, sFlt1).

Studies also demonstrated that, for a patient presenting a placental vascular pathology, the rate of PlGF is decreased and conversely for the rate of sFlt1. Studies show that the duration of the pregnancy, of a patient presenting a placentary vascular pathology, is correlated at the rate of these markers.

There is at present no reliable predictive examination to estimate the arisen of severe complications for a patient presenting a placental vascular pathology. The purpose of the study will to estimate the relevance of the serum markers sFlt1 and PlGF to predict the arisen of severe complications for these patients.

ELIGIBILITY:
Inclusion Criteria:

* pregnant woman with a diagnosis of placental vascular disease (gestational hypertension, preeclampsia, IUGR)

Exclusion Criteria:

* patient who refuses the obstetric follow-up

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All pregnant women with a diagnosis of placental vascular disease during the third trimester
Sampling Method: Non-Probability Sample
Enrollment: 233 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Arisen of a maternal and/or fetal severe complication | during the pregnancy from 24 weeks of gestation until delivery
  The severe maternal complication are : placental abruption, HELLP syndrome, Lung acute oedema ; eclampsia, maternal death.
  The fetal severe complications are : intrauterine grow retardation, fetal demise.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe DOCHE, Study Director — Centre Hospitalier Metropole Savoie
Locations (7):
- France (7):
  - CHMetropoleSavoie, Chambéry, Savoie
  - CHU de Brest, Brest
  - Centre Hospitalier Alpes Léman, Contamine-sur-Arve
  - Groupe Hospitalier du Havre, Le Havre
  - CHU de Limoges, Limoges
  - Centre Hospitalier Annecy Genevois, Metz-Tessy
  - Hôpitaux du Léman, Thonon-les-Bains

IPD SHARING:
Plan to Share IPD: No